CLINICAL TRIAL: NCT02911246
Title: Evaluation Report of the Urea / Urine Creatinine as a Marker of Nutritional Status Predictive of ICU Care Associated Infections
Acronym: UREA
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC13_0353
Record Dates: First submitted 2016-09-12; First posted 2016-09-22 (Estimated); Last update posted 2016-09-23 (Estimated); Status verified 2016-09

CONDITIONS: Brain Injury; Malnutrition
MeSH Terms: conditions — Brain Injuries; Malnutrition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Malnutrition is defined by an energy supply deficit, protein, macro-molecules or micro-nutrients, resulting from an imbalance between nutrient intakes and metabolic needs of the body. It concerns 40 to 60% of patients upon entry into resuscitation and influences their prognosis. Studies over the past decade have shown that nutritional deficiency increases the morbidity and mortality in intensive care.

Several clinical and biological parameters were evaluated as markers of malnutrition, including the ratio of urea / urine creatinine.

The report would identify patients in a state of malnutrition, to optimize their nutritional care.

This setting is easy to obtain in all patients by simple urine collection unlike other clinical and biological criteria of resuscitation malnutrition assessment.

This ratio of urea / urien creatinine would optimize energy intake of critically ill patients, for which nutritional management methods are widely debated.

DETAILED DESCRIPTION:
At present, many clinical studies have shown a link between malnutrition and infectious complications in intensive care particularly because of immune disorders.

Many studies testing different nutritional strategies used as the main criterion infectious complications.

So this is a robust standard, well documented in the literature as a reflection of malnutrition in intensive care, and we also want to use in our study.

In a pilot study in the surgical ICU of the Hotel-Dieu report the urea / creatinine urine as a biomarker of poor outcome of nutritional status in the ICU seems extremely discriminating in predicting the existence of nosocomial infection.

Furthermore the kinetics of the relationship between the intake and the 5th day of resuscitation, also appears to be relevant in predicting the occurrence of nosocomial infection.

Surgical ICU of the Hotel-Dieu proposes to conduct a multicenter study to confirm the relationship between the ratio of urea / creatinine urine, malnutrition marker, and nosocomial infections (NI) in intensive care.

Primary objective:

To evaluate the predictability of the ratio of urea / creatinine urinary J5 on the occurrence of nosocomial infection in intensive care.

ELIGIBILITY:
Inclusion Criteria:

* 18 or more
* Admission in ICU
* Estimated length of stay superior to 5 days

Exclusion Criteria:

* pathologies modifying the ratio of urea / urine creatinine: end stage renal disease ( creatinine clearance less than 15 mL / min), Gastrointestinal bleeding, Right ventricular failure

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized in ICU for severe brain injury
Sampling Method: Non-Probability Sample
Enrollment: 309 (Actual)
Dates: Start 2014-12; Primary Completion 2014-12 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Number of infections related to care during stay in intensive care unit | 5 days after admission
  Six infections assessed are:
  1. Nosocomial pneumonia and tracheobronchitis
  2. urinary infection
  3. surgical site infection
  4. bacteraemia
  5. intra-abdominal infection
  6. Infection of the central nervous system

CONTACTS AND LOCATIONS:
Overall Officials: Karim Asehnoune, MD PhD, Principal Investigator — Nantes University Hospital

IPD SHARING:
Plan to Share IPD: Undecided